CLINICAL TRIAL: NCT05919329
Title: Modulation of PSMA Expression in Castration Sensitive and Castration Resistant Prostate Cancer in Response to Hormonal Therapy
Brief Title: Evaluation of the Change in PSMA Expression in Prostate Cancer in Response to Hormonal Therapy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Nadine Mallak, MD, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00025799; NCI-2023-06184 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Castration Resistant Prostate Cancer; Castration Sensitive Prostate Cancer; Prostate Adenocarcinoma
MeSH Terms: interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid; Magnetic Resonance Spectroscopy; Specimen Handling

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1: CRPC (Experimental): Patients with CRPC will receive 18F-DCFPyL PET prior to start of therapy (standard of care), then again 8 days and 28 days after initiation of hormonal therapy.
  Interventions: Drug: Piflufolastat; Procedure: PSMA PET/CT Scan; Procedure: PSMA PET/MRI scan; Procedure: Biospecimen Collection; Other: Electronic Health Record Review
- Cohort 2: CSPC (Experimental): Patients with CSPC will receive 18F-DCFPyL PET prior to start of therapy (standard of care), then again 8 days and 28 days after initiation of hormonal therapy.
  Interventions: Drug: Piflufolastat; Procedure: PSMA PET/CT Scan; Procedure: PSMA PET/MRI scan; Procedure: Biospecimen Collection; Other: Electronic Health Record Review

INTERVENTIONS:
Drug: Piflufolastat — Given IV
  Other Names: Piflufolastat F-18; Pylarify; 18F-DCFPyL; Fluorine F 18 DCFPyL
Procedure: PSMA PET/CT Scan — Undergo PSMA PET/CT
  Other Names: Prostate-Specific Membrane Antigen PET/CT; PSMA PET/CT; PSMA-Positron emission tomography/CT
Procedure: PSMA PET/MRI scan — Undergo PET/MRI
  Other Names: Prostate-Specific Membrane Antigen PET/MRI; PSMA PET/MR; PSMA-Positron emission tomography/magnetic resonance imaging
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Specimen Collection; Lab draw
Other: Electronic Health Record Review — Ancillary studies

SUMMARY:
This clinical trial investigates the change in prostate-specific membrane antigen (PSMA) expression in response to hormonal therapy in both, Castration Sensitive Prostate Cancer (CSPC) and Castration Resistant Prostate Cancer (CRPC), and whether this change in PSMA expression changes tumor staging after therapy initiation. Understanding these effects can help define the best timing to perform the PSMA positron emission tomography (PET) relative to the start of therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the early effects (at day 8) of hormonal therapy on PSMA modulation in patients with castration sensitive prostate cancer (CSPC) and castration resistant prostate cancer (CRPC)

SECONDARY OBJECTIVES:

I. To evaluate the effects of hormonal therapy on PSMA modulation at day 28 post-therapy in patients with CSPC and CRPC

II. To evaluate whether the change in PSMA modulation after hormonal therapy initiation changes the tumor staging on PSMA PET as defined by the PROMISE V2 criteria.

EXPLORATORY OBJECTIVES:

I. To assess whether the initial change in PSMA modulation in response to hormonal therapy holds prognostic implications

II. To assess for potential correlation between the early change in PSMA modulation and tumor characteristics such as Gleason score, and site of disease.

III. To assess whether the baseline level of PSMA uptake holds prognostic implications in response to hormonal therapy

OUTLINE:

Patients will be divided (non-randomized) into 2 groups (CRPC or CSPC) and receive PSMA PET prior to start of therapy (standard of care), then again 8 days and 28 days after initiation of hormonal therapy.

Participants will be followed for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant or legally authorized representative (LAR) must provide written informed consent before any study-specific procedures or interventions are performed.
* Participants must have confirmed prostate adenocarcinoma, histologically, or by combined imaging and biochemical markers.
* Age >= 18 years. Given the nature of the disease in question, only men will be included. Members of all races and ethnic groups will be included.
* Participants must have sites of prostate cancer showing uptake on an initial PSMA PET scan.
* Participants are planned to receive hormonal therapy within eight weeks of the initial PSMA PET. The hormonal therapy agents include:

  * For CSPC: GnRH agonists, GnRH antagonists, first-generation antiandrogen (e.g. bicalutamide), or androgen receptor (AR)-targeted agent (e.g. Abiraterone, Enzalutamide, Apalutamide, Darolutamide)
  * For CRPC: this group of patients are typically on continuous ADT (GnRH agonists or antagonists), which will be continued, and the hormonal therapy they will be started on is an androgen receptor (AR)-targeted agent (e.g. Abiraterone, Enzalutamide, Apalutamide, Darolutamide)
* Life expectancy > 3 months.
* Cohort 1: Castration resistant prostate cancer with rising PSA (confirmed by two PSA values at least 1 week apart), testosterone < 50 ng/dL, on continuous ADT at least 4 months, no AR targeted agent in the prior 4 months.
* Cohort 2: Castration sensitive prostate cancer with no ADT or AR targeted agents use in the past 12 months, testosterone >50 ng/dL

Exclusion Criteria:

* Uncontrolled serious infection.
* Intercurrent illness or condition that would limit compliance with study requirements.
* Participants who have undergone any cancer treatment other than the hormonal therapy (systemic or radiation therapy) or who have started any supplements or herbal medications intended to treat cancer between the baseline PSMA PET and PSMA PET at day 28.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in maximum standardized uptake value (SUVmax) on post-therapy initiation PSMA PET (8 ± 2 days) compared to baseline. | Baseline PSMA PET up to 8 days after therapy initiation
  Evaluate the change in SUVmax between baseline and Day 8 using a paired t-test to determine how hormonal therapy affects the PSMA modulation.

SECONDARY OUTCOMES:
Change in SUVmax on post-therapy initiation PSMA PET (28 ± 3 days) compared to baseline. | Baseline PSMA PET up to 28 days after therapy initiation
  Evaluate the change in SUVmax between baseline and Day 28 using a paired t-test to determine how hormonal therapy affects the PSMA modulation.
Number of patients in whom the tumor staging changed on PSMA PET scans obtained post-therapy initiation relative to baseline PET scan | Baseline PSMA PET up to 28 days after therapy initiation

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Mallak, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States